CLINICAL TRIAL: NCT01639612
Title: A Pilot Safety Study of the Administration of Bone Marrow Derived Stem Cells (ALD-451) in WHO Grade IV Malignant Glioma
Brief Title: Pilot Study of Bone Marrow/Stem Cells in Grade IV Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Henry Friedman (Other)
Responsible Party: Sponsor-Investigator, Henry Friedman, Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00031192
Record Dates: First submitted 2012-06-28; First posted 2012-07-13 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Grade IV Malignant Glioma
Keywords: Stem Cell; Grade IV Malignant Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ALD-451 (Experimental): Autologous bone marrow derived ALD-451 cells administered intravenously following surgery, radiation therapy and temozolomide
  Interventions: Biological: ALD-451

INTERVENTIONS:
Biological: ALD-451 — ALD-451 iv

SUMMARY:
1. Purpose of the Study - This protocol aims to demonstrate the feasibility and safety of autologous ALD-451 cells administered intravenously in World Health Organization (WHO) grade IV malignant glioma patients following surgery, radiation therapy and temozolomide; as well as to obtain an initial description of the effects of ALD-451 cells on neuro-cognition allowing the design of a subsequent phase 2 trial of this intervention in patients with malignant glioma. The primary objective of this study is to demonstrate the safety of intravenously administered autologous bone marrow derived ALD-451 cells in the brain following surgery, radiation therapy and temozolomide in patients with WHO grade IV malignant glioma. The secondary objective of this study is to determine the recovery of ALD-451 from bone marrow of patients following radiation therapy and temozolomide. The exploratory objective of this study is to determine if intravenous administration of autologous ALD-451 cells following surgery, radiation therapy and temozolomide in WHO grade IV malignant glioma patients may have an effect on subsequent deterioration of neurocognition and patient-reported outcomes.

DETAILED DESCRIPTION:
This is a pilot, open label study in which eligible subjects will undergo surgery, radiation therapy, Temozolomide, bone marrow harvest, MRIs, and intravenous infusion of ALD-451. The subjects will be followed via the safety and efficacy procedures completed during visits over 12 months.

Two to 8 weeks following gross total resection (GTR), patients with WHO grade IV malignant glioma that have agreed to participate in the study by signing the informed consent will undergo screening procedures to determine eligibility. Once enrolled on the study, baseline neurocognitive testing will be performed. Two to 8 weeks after enrolled subjects have completed the 6 -6 ½ weeks of radiation therapy and daily temozolomide, subjects will have their bone marrow harvested by undergoing a bone marrow aspiration with 160 (+/-20) mL of bone marrow collected from the iliac crest (one to 2 days after the patient has been re-assessed for continued eligibility).

The sample will be transported to the Robertson CT2 GMP Facility where ALD-451 will be manufactured and the ALD-451 product returned to the Investigational Chemotherapy Services for infusion. A small aliquot of ALD-451 will be taken from the starting bone marrow, de-identified, labeled with the manufacturing lot number, and stored at Duke University for the duration of the trial to support ongoing studies determining potency of the product. For all ALD-451 products, a retained aliquot that is the equivalent of 10 mls of the starting bone marrow will be cryopreserved and stored in the vapor phase of liquid nitrogen. Harvest of 160 mL of subject bone marrow will allow for retains without excessive reduction in the anticipated ALDHbr dose. These frozen retains will be used for product characterization and development of a potency assay. These aliquots will not be used for any other purposes and any remaining aliquots will be destroyed at the time of Biologics License Application (BLA) approval.

Two - four days after having bone marrow harvested for ALDHbr cells, ALD-451 will be administered through a peripheral IV, up to 1 hour. This will be followed by 4 hours of IV fluids and observation. Normal Saline will be used as the IV fluids and will be initiated a few minutes before the administration of ALD-451. The bag within which ALD-451 will be received will be flushed once with 10 ml of Normal Saline and the fluid obtained after flushing the bag will be administered to the patient, to assure that the investigators have reinfused in the patient the vast majority of the ALD-451 present in the bag.

Temozolomide will be reinitiated four weeks after completion of radiation therapy and daily Temozolomide (at least two weeks after ALD-451 infusion). Temozolomide will be dosed at 150 mg/m2 orally on days 1-5 of a 28-day cycle for the first cycle and 200 mg/m2 orally for the following 11 cycles. Patients will receive a total of 12 cycles of Temozolomide following completion of radiation therapy.

Neurocognitive testing and patient-reported outcomes will be obtained at study enrollment, two weeks after completion of radiation therapy and temozolomide and after six and twelve cycles of temozolomide.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria are as follows:

1. Newly diagnosed patients with histologically proven supratentorial primary WHO grade IV malignant glioma (glioblastoma or gliosarcoma) with gross total resection (less than 1 cm of residual disease in the maximal diameter).
2. Age ≥ 18 years of age.
3. Karnofsky Performance Status ≥ 60%.
4. Adequate renal function, defined as creatinine ≤ 1.3 mg/dL (μmol/L).
5. Adequate serum chemistry parameters. Total bilirubin ≤ 1.5 x upper limit of normal (ULN) and aspartate aminotransferase (AST) ≤ 2.5 X the ULN.
6. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
7. Women of childbearing potential must have a negative serum pregnancy test in the 48 hours prior to enrollment.
8. Men and women of reproductive potential must agree to use an effective contraceptive method including one of the following: surgical sterilization (tubal ligation for women or vasectomy for men); approved hormonal contraceptives (such as birth control pills, patches, implants or injections); barrier methods (such as condom or diaphragm) used with a spermicidal cream or an intrauterine device (IUD). Contraceptive measures such as Plan B ™, sold for emergency use after unprotected sex, are not acceptable methods for routine use.
9. Is able to provide bone marrow sample from iliac crest.
10. Is able to return for dosing two days post bone marrow harvest for infusion at Duke University.
11. Is able to interrupt anticoagulation (if applicable) for bone marrow harvest and dosing procedures.
12. Patient willing to undergo external beam radiation therapy and chemotherapy with Temozolomide at Duke University Medical Center and stay four hours post infusion of ALD-451.
13. Patient must give written informed consent prior to any study-specific procedures being implemented.
14. Is a good candidate for the trial, in the opinion of the investigator.

Exclusion Criteria:

Exclusion Criteria are as follows:

1. Primary WHO grade IV malignant glioma (glioblastoma or gliosarcoma) with an infratentorial lesion or involvement of the spinal cord.
2. Patients with more than 1 cm of residual tumor in the maximal diameter at the post surgery MRI.
3. Pregnant or lactating females.
4. Women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception.
5. Prior chemotherapy, immunotherapy, biologic therapy, radiation therapy, radioimmunotherapy, hormonal therapy, or experimental therapy for brain tumor. Prior or active corticosteroid therapy is permitted to control neurologic symptoms due to intracranial edema.
6. History of severe allergic reaction to contrast media.
7. Any serious medical condition or psychiatric illness unresponsive to medical intervention.
8. Prior malignancy if active treatment was required during the previous 5 years except for adequately treated basal cell or squamous cell skin cancer and in situ uterine cervical cancer.
9. Myocardial infarction in the past 3 months.
10. Mechanical heart valve.
11. Medical history or neurological pathology that prevents neurocognitive testing and prescribed patient outcome reporting.
12. Any concurrent illness or condition that in the opinion of the investigator might interfere with treatment or evaluation of safety and/or efficacy.
13. Current or recent history of alcohol or drug abuse.
14. Known history of infection with HIV or hepatitis.
15. Active systemic infection requiring IV antibiotics.
16. Subjects currently receiving restricted concomitant medications.
17. Any previous or current treatment with angiogenic growth factors, cytokines, gene therapy or stem cell therapy.
18. Unable to return for follow up visits for clinical evaluation, safety evaluation, laboratory studies, or MRI evaluation.
19. Inability to undergo an MRI.
20. Hemoglobin < 10g/dl.
21. Platelet counts of < 100,000 or > 700,000 at screening.
22. Hypertension with systolic BP ≥ 150mmHg or diastolic BP≥95 mmHg despite adequate anti-hypertensive treatment.
23. Patients treated on any other therapeutic clinical protocols within 30 days prior to study entry or during participation in the study.
24. Any previous or current treatment with stem cell therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-06; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with unacceptable toxicity | 12 months after study drug administration
  Number of patients with irreversible Grade 3 or greater central nervous system (CNS) toxicity or Grade 3 or greater non-hematologic toxicity if attributable to ALD -451

SECONDARY OUTCOMES:
Number of ALD-451 cells recovered from bone marrow of patients following radiation therapy and chemotherapy | Baseline to 48 weeks
Neurocognition and patient-reported outcomes following ALD-451 | Baseline to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States